CLINICAL TRIAL: NCT00000757
Title: A Phase I Multicenter Trial to Evaluate the Safety and Immunogenicity of HIV-1 Recombinant Envelope Glycoprotein gp160
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 003A; 10541 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; HIV-1; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To evaluate the safety and immune response to 160 mcg HIV-1 recombinant envelope glycoprotein gp160. To evaluate the duration of antibody response and its relationship to dose and frequency of inoculation.

Evaluation of previous patients who received doses of 40 or 80 mcg gp160 vaccine indicate that, although serum anti-gp160 antibody responses were detected, the level and duration of those responses were limited. A preliminary observation suggests that weak functional antibody responses may develop following the 18 month booster of 40 or 80 mcg; therefore, a dose of gp160 vaccine having potentially greater immunogenicity is of particular interest.

DETAILED DESCRIPTION:
Evaluation of previous patients who received doses of 40 or 80 mcg gp160 vaccine indicate that, although serum anti-gp160 antibody responses were detected, the level and duration of those responses were limited. A preliminary observation suggests that weak functional antibody responses may develop following the 18 month booster of 40 or 80 mcg; therefore, a dose of gp160 vaccine having potentially greater immunogenicity is of particular interest.

Healthy volunteers are injected on days 0, 30, 180, and 365 with either 160 mcg gp160 vaccine (20 volunteers) or an alum placebo preparation (10 volunteers).

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative for HIV infection by ELISA and Western blot (i.e., no reactivity at gp160, gp120, gp41, or p24).
* T4 count >= 800 cells/mm3.
* Normal chest x-ray and urinalysis.
* Negative hepatitis B surface antigen.
* Negative HIV p24 antigen test.
* Normal skin reactivity by Merieux test.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive PPD.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease).

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or use of immunosuppressive medications.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.

Prior Treatment:

Excluded:

* Prior blood transfusions or cryoprecipitates within the past 6 months.

Identifiable high-risk behavior for HIV infection (as determined by prescreening questions designed to identify risk factors for HIV infection), including:

* Any history of IV drug use.
* Syphilis, gonorrhea, or any other sexually transmitted diseases (including chlamydia or pelvic inflammatory disease) in the past 6 months.
* More than two sexual partners, or sexual contact with a high-risk partner, in the past 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Study Completion 1992-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair; Clements ML, Study Chair; Couch R, Study Chair; Dolin R, Study Chair; Levine M, Study Chair; Wright P, Study Chair
Locations (1):
- St. Louis Univ. School of Medicine AVEG, St Louis, Missouri, United States

REFERENCES:
- [Background] Keefer MC, Wolff M, Gorse GJ, Graham BS, Corey L, Clements-Mann ML, Verani-Ketter N, Erb S, Smith CM, Belshe RB, Wagner LJ, McElrath MJ, Schwartz DH, Fast P. Safety profile of phase I and II preventive HIV type 1 envelope vaccination: experience of the NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1997 Sep 20;13(14):1163-77. doi: 10.1089/aid.1997.13.1163. PMID 9310283
- [Background] Keefer MC, Graham BS, Belshe RB, Schwartz D, Corey L, Bolognesi DP, Stablein DM, Montefiori DC, McElrath MJ, Clements ML, et al. Studies of high doses of a human immunodeficiency virus type 1 recombinant glycoprotein 160 candidate vaccine in HIV type 1-seronegative humans. The AIDS Vaccine Clinical Trials Network. AIDS Res Hum Retroviruses. 1994 Dec;10(12):1713-23. doi: 10.1089/aid.1994.10.1713. PMID 7888231